CLINICAL TRIAL: NCT00037193
Title: Acute Regulation of Parathyroid Hormone by Dietary Phosphate
Status: Completed | Type: Observational
Sponsor: National Center for Research Resources (NCRR) (NIH)
Other Study IDs: NCRR-M01RR00036-0855
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Secondary Hyperparathyroidism
MeSH Terms: conditions — Hyperparathyroidism, Secondary

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Patients with end stage renal disease often have secondary hyperparathyroidism due to high phosphorus and low calcium levels in the blood. Preliminary animal studies and our initial human study indicate that the parathyroid hormone levels may change quickly based on the ingestion of phosphorus, prior to any change in the blood levels of calcium or phosphorus. This follow-up study will attempt to determine if the effect is independent of an increase in the blood glucose level. If so, this would suggest an as yet unidentified gastrointestinal receptor that mediates parathyroid hormone levels. This may affect the timing of administration and the type of phosphate binder used in treating patients with secondary hyperparathyroidism. The knowledge that parathyroid hormone levels can change acutely may also affect the recommended timing of blood samples

DETAILED DESCRIPTION:
This study is observational and no drugs or other interventions will be used. The population targeted in this study will be adult patients already on chronic hemodialysis with a diagnosis of secondary hyperparathyroidism. Experimental design will involve the use of a glucose clamp to maintain a constant, mild increase in blood glucose levels. Frequent, scheduled lab tests will be obtained during the period of hyperglycemia to evaluate phosphorous, calcium, and glucose levels and the relationship of any change in their values to changes in the parathyroid hormone level. The primary outcome will be to evaluate for any change in the parathyroid hormone level in the presence of hyperglycemia and to compare these results to that of our initial study

ELIGIBILITY:
1. Patients 21 years of age or older
2. Receiving treatment with hemodialysis for at least 90 days.
3. Serum parathyroid hormone level greater than 200 pg/ml
4. Serum phosphorus level greater than 4 mg/dl

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Washington University Medical School, St Louis, Missouri, United States